CLINICAL TRIAL: NCT01772186
Title: Freezing of Gait Correction and Fall Prevention in People With Parkinson's Disease: Developing and Application of a Real-time Somatosensory Stimulation System
Brief Title: Freezing of Gait Correction and Fall Prevention: Developing a Real-time Somatosensory Stimulation System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Ruey-Meei Wu, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201112158DIB
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: Parkinson Disease
Keywords: Freezing of gait; Parkinson's disease; Somatosensory stimulation; Fall prevention
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Without real-time somatosensory cue (No Intervention): Parkinson patients wear the somatosensory stimulation system but not receive the real-time somatosensory cue during freezing-of-gait episodes.
- With real-time somatosensory cue (Experimental): Parkinson patients wear the somatosensory stimulation system and receive the real-time somatosensory cue during freezing-of-gait episodes.
  Interventions: Device: Real-time somatosensory cue

INTERVENTIONS:
Device: Real-time somatosensory cue — A novel sensory cue proposed in this study, which designed to facilitate weight shift during freezing-of-gait episodes. This sensory cue is controlled by the real-time analysis of gait pattern, and given only when freezing-of-gait detected.
  Arms: With real-time somatosensory cue

SUMMARY:
Background and purpose: Freezing of gait (FOG) is one of the most disabling motor symptoms in people with Parkinson's disease (PD), and closely associates with postural instability and fall. Previous studies had shown that somatosensory stimulation could induce weight shift, and this is probably helpful for gait reinitiation. Therefore, the investogators propose a two-year project to develop a wearable device, the somatosensory stimulation system (SSS), which monitors gait real-time and provide somatosensory stimulation once FOG episodes detected. And the investigators test the effects of this SSS device on FOG, fall, and walking function.

Methods: The first-year study is to build and validate this wearable SSS device. The customized device has sensor part and stimulator part; the former is an inertial sensor module to detect FOG episodes, and the latter is a microvibrator-embedded insole to facilitate weight shift and gait reinitiation. To validate the device, patients with FOG are recruited and conduct FOG-provoking tasks during their medication "OFF" or "late On" state in a laboratory setting. The investigators test if the SSS device could facilitate lateral weight shift and help gait reinitiation, as well as the reliability. The second-year study is to test if the SSS device stands a long-term, daily wearing basis, and to evaluate its effect on FOG, fall, and walking function. The investigators recruit PD patients with FOG, and randomly assign them into the experimental and control groups. Both groups wear the SSS device during the daytime for ten weeks, and the stimulator part is turned on during the first six weeks (intervention phase) only in the experimental group. The stimulator part is then kept off during the last four weeks (follow-up phase) in both groups. The effect of the SSS device is evaluated by the outcomes including FOG severity, fall and walking function, which are measured prior/after the intervention phase and after the follow-up phase.

Clinical relevance: This project tempts to combine real-time gait analysis with somatosensory-induced postural readjustment, and using this novel approach to improve FOG and fall in people with PD. The results of this projects might also provide an objective, long-term assessment tool to measure the FOG phenomenon for clinical and research fields.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinsonian with Hoehn-Yahr score between 2 to 4
* Suffering freezing-of-gait in the recent week
* Able to walk unassisted over 30 meters in medication OFF period

Exclusion Criteria:

* Non-idiopathic Parkinsonian
* Comorbid with uncontrolled neurological, cardiovascular and orthopedic diseases that might affect balance and mobility
* Impaired cognitive function
* Abnormal plantar sensory function
* Abnormal coagulation function

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Reliability of the somatosensory stimulation system | 2 weeks
  The reliability of the somatosensory stimulation system in detecting freezing-of-gait episodes during gait.
Validity of the somatosensory stimulation system | 2 weeks
  If the somatosensory stimulation system can facilitate weight shift and help gait reinitiation during freezing-of-gait.
Fall prevention | 10 weeks
  If the somatosensory stimulation system can reduce the incidence of fall in people with Parkinson disease.

CONTACTS AND LOCATIONS:
Overall Officials: Ruey-Meei Wu, Professor, Principal Investigator — Department of Neurology, National Taiwan University Hospital, College of Medicine, National Taiwan University, Taipei, Taiwan; Kwan-Hwa Lin, Professor, Principal Investigator — Department of Physical Therapy, Tzu Chi University, Hualien, Taiwan
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei, Taiwan
  - National Taiwan University Hospital, Taipei